CLINICAL TRIAL: NCT01657981
Title: An Open Label Study to Evaluate the Pharmacokinetics of YM150 After a Single Oral Dose of C14-labeled YM150 in Healthy Male Subjects
Brief Title: A Study to Find Out How YM150 is Absorbed Into and Eliminated From the Body in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 150-CL-015; 2006-001968-22 (EudraCT Number)
Record Dates: First submitted 2012-07-10; First posted 2012-08-06 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2012-08

CONDITIONS: Pharmacokinetics; Healthy Male Subjects
Keywords: Pharmacokinetics; Phase 1; 14C-labeled
MeSH Terms: interventions — darexaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm 1 (Experimental)
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — 14C-labeled YM150, oral solution
  Other Names: darexaban

SUMMARY:
The study aims to observe how YM150 was absorbed, distributed and excreted after dosing with a radio labeled drinking solution.

DETAILED DESCRIPTION:
Healthy male subjects are admitted on Day 0. Subjects receive a single oral dose of 14C-labeled YM150 in the morning of Day 1 and remain in the unit for 7 days (6 nights). Blood, plasma, urine and feces samples are collected until 120 hrs after dosing for analysis of 14C-labeled radioactivity, YM150, YM-222714 and other metabolites. Expired air is collected as well for assessment of 14C-radioactivity.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60 and 100 kg and Body Mass Index between 18 and 30 kg/m2

Exclusion Criteria:

* Known or suspected hypersensitivity to YM150 or any of the constituents of the formulations used
* History of and/or any sign or symptom indicating current abnormal hemostasis or blood dyscrasia, including but not limited to neutropenia, thrombocytopenia, thrombocytopathy, thromboasthenia, hemophilia, Von Willebrand's disease, and vascular purpura, bleeding gums or frequent nose bleeding
* Family history of congenital vascular malformation (e.g. Marfan's Syndrome) and/or bleeding disorder (e.g. hemophilia, Von Willebrand's disease, Christmas disease)
* History of peptic ulcer or of any other organic lesion susceptible to bleeding
* Prothrombin time (PT) or Activated partial thromboplastin time (aPTT) at the screening visit outside the normal range
* Any surgical intervention (including tooth extraction) or trauma within the last 3 months preceding the start of the study
* Any clinically significant history of asthma, eczema, any other clinically significant allergic condition or previous severe hypersensitivity to any other drug
* Any clinically significant upper gastro-intestinal symptoms likely to interfere with the absorption of the drug
* History or presence of any cardiovascular disease or disorder
* History of a clinically significant ECG abnormality
* Any clinically relevant history of other disease or disorder - gastrointestinal, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic
* Any clinically significant abnormality following the Investigator's review of the pre-study physical examination, ECG, and clinical laboratory tests
* Abnormal heart rate and blood pressure measurements at the screening visit as follows: heart rate <40 or >90 bpm; mean systolic blood pressure <95 or >160 mmHg; mean diastolic blood pressure <40 or >95 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min)
* Regular use of any prescribed or OTC drugs (including vitamins and herbal remedies) in the 4 weeks prior to admission to the clinical unit OR any use of such drugs in the 2 weeks prior to admission to the clinical unit
* History of drug abuse at any time, OR any use of drugs of abuse within 3 months prior to admission to the clinical unit
* Participation in any clinical study within 3 months, or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study
* History of drinking more than 21 units of alcohol per week (1 unit = 270 ml of beer or 40 ml of spirits or 125 ml of wine) within 3 months prior to admission to the clinical unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit
* Subject, who is anti-HAV (IgM), anti-HCV, HBsAg or HIV-1 or -2 positive
* Donation of blood (>400 ml) or blood products within 3 months prior to admission to the clinical unit or plasmapheresis within 4 weeks prior to admission to the clinical unit
* Exposure to radiation for diagnostic reasons (except dental X-rays and plain X-rays of thorax and bony skeleton (excluding spinal column)), during work or during participation in a clinical study in the previous year

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of 14C-labeled YM150 assessed by whole blood, plasma, urine, feces and expired air concentrations | Day 1 - Day 6
  AUCinf (Amount excreted in urine extrapolated until infinity), AUClast (Amount excreted in urine until last sample), Cmax (Maximum concentration), tmax (Time to attain maximum concentration), tlag (Absorption lag time) and t1/2 (Apparent terminal elimination half-life). Excretion rate and cumulative excretion of radioactivity in urine, feces and expired air.
Pharmacokinetics of YM150 and metabolites assessed by plasma and urine concentrations | Day 1 - Day 6
  - AUCinf, AUClast, Cmax, tmax, tlag and t1/2. In urine - amount excreted in urine, CLR (Renal clearance) and % of dose excreted.

SECONDARY OUTCOMES:
Identification of the metabolic profile of YM150 in human plasma, urine and feces | 0 - 2 hours Day 1
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | Day 1 - 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- PRA International EDS NL, Zuidlaren, Netherlands